CLINICAL TRIAL: NCT01391949
Title: UCFit Pedaling Exercises to Limit Disability in the Outpatient Setting
Brief Title: Pedaling Exercises for Disability and Activity Limitations
Acronym: PEDAL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Bruce H. Dobkin, Professor of Neurology, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11-001404
Record Dates: First submitted 2011-07-11; First posted 2011-07-12 (Estimated); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Stroke
Keywords: disability; walking; feedback; exercise
MeSH Terms: conditions — Stroke; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Detailed feedback (Experimental): Subjects will pedal on the UCFit with a goal of 30 total minutes of daily exercise.
  Interventions: Behavioral: Detailed feedback
- Basic feedback (Active Comparator): Subjects will pedal on the UCFit with a goal of 30 total minutes of daily exercise.
  Interventions: Behavioral: Basic feedback

INTERVENTIONS:
Behavioral: Detailed feedback — Once a week subjects will receive feedback about the total time spent cycling and walking in the previous week. Subjects in this intervention group will also receive feedback about average cycling speed, distance pedaled, average walking speed, and distance walked in the previous week.
  Arms: Detailed feedback
Behavioral: Basic feedback — Once a week subjects will receive feedback about total time spent cycling and walking in the previous week.
  Arms: Basic feedback

SUMMARY:
This purpose of this study is to determine the effect of different levels of feedback on participation in a home exercise regimen and the amount of walking performed by patients recently discharged from the acute rehabilitation setting.

DETAILED DESCRIPTION:
The UCFit (University of California's U Cycle to Fitness) device is a standard commercial arm and leg restorator modified to collect pedaling data and to transmit it wirelessly to a central database, allowing for remote exercise monitoring. In this study, patients with stroke will perform pedaling exercise on the UCFit device prior to and then for a period of twelve weeks after discharge to home from inpatient rehabilitation. Differing levels of feedback will be provided to study subjects and corresponding changes in the amount of pedaling and walking performed will be identified. The results of this study will offer insight into the activity levels of disabled persons in their home environments. Furthermore, it will help in the identification of strategies that can increase activity levels in the critical period after discharge to home.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of stroke
* no major contraindications to participating in light-to-moderate exertion
* able to follow and retain verbal directions to carry out simple lower extremity repetitive exercises
* planned discharge to home with family available to assist

Exclusion Criteria:

* pre-morbid limitations in walking related to another medical disease
* body mass index >30
* fractures or contractures that prevent use of an extremity for pedaling
* impairment in cognition that precludes a full understanding of the risks and benefits of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2011-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Walking speed | three months
  Fastest safe walking speed over 10 meters

SECONDARY OUTCOMES:
Distance walked in 3 minutes | three months
  Distance walked at fastest safe speed over 3 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Dorsch, MD, Principal Investigator — University of California, Los Angeles; Bruce Dobkin, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States